CLINICAL TRIAL: NCT07058012
Title: A Phase II Platform Study to Evaluate Treatment With Cemiplimab Monotherapy or Cemiplimab Plus Fianlimab and Other Novel Combinations in Patients With Colorectal Cancer With Minimal Residual Disease Following Definitive Surgery and Chemotherapy
Brief Title: A Phase II Platform Study to Evaluate Treatment With Cemiplimab Monotherapy or Cemiplimab Plus Fianlimab or Other Novel Combinations in Patients With Colorectal Cancer With Minimal Residual Disease Following Definitive Surgery and Chemotherapy (EMPIRE)
Acronym: EMPIRE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NSABP FC-13
Record Dates: First submitted 2025-03-06; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Arm 1 (Active Comparator): cemiplimab
  Interventions: Drug: Cemiplimab; Other: ctDNA testing
- Arm 2 (Active Comparator): cemiplimab plus fianlimab
  Interventions: Drug: cemiplimab plus fianlimab; Other: ctDNA testing
- Arm 3 (Experimental): cemiplimab plus REGN7075
  Interventions: Drug: cemiplimab + REGN7075; Other: ctDNA testing

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab 350mg intravenously
  Arms: Arm 1
Drug: cemiplimab plus fianlimab — Cemiplimab 350mg + Fianlimab 1600mg intravenously
  Arms: Arm 2
Drug: cemiplimab + REGN7075 — Cemiplimab 350mg + REGN7075 2700mg intravenously
  Arms: Arm 3
Other: ctDNA testing — Eligible patients using results for ctDNA-positivity as obtained from a commercial assay run in any CLIA-certified lab will proceed to enrollment and begin treatment. All patients will have confirmation of ctDNA-positivity via the Signatera^TM assay (Clinical Trial Assay), but treatment may proceed while awaiting confirmatory results.
  Other Names: Signatera; Other

SUMMARY:
The NSABP FC-13 study is being done to determine if using immunotherapies alone or in combination with other drugs will delay or prevent colorectal cancer from coming back in patients with colorectal cancer who are ctDNA-positive after their treatment. Immunotherapeutic drugs (immunotherapies) act on different proteins on the surface of cells of the immune system and trigger the immune system to destroy cancer cells. The drugs being studied in NSABP FC-13 are cemiplimab, fianlimab, and REGN7075.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and, prior to beginning specific study procedures, must have signed and dated appropriate Institutional Review Board (IRB) -approved consent forms that conform to federal and institutional guidelines for study treatment.
* Patients must be greater than or equal to18 years old.
* The ECOG performance status must be 0-1.
* Patients must have confirmed histologic and pathologic stage II/III colon, stage II/III rectal, or oligometastatic stage IV colorectal adenocarcinoma (per AJCC 8th edition).
* There must be documentation by CT scan with contrast that the patient has no definitive evidence of metastatic disease including assessment of chest, abdomen, and pelvis at the time of study enrollment
* All patients must have had a complete (R0) resection of their primary tumor and oligometastatic disease if present AND at least 3 months of a standard systemic chemotherapy regimen (e.g., FOLFOX or CAPOX or fluoropyrimidine monotherapy). This includes either adjuvant chemotherapy for colon cancer or perioperative (adjuvant or neoadjuvant) chemotherapy for rectal cancer or oligometastatic colon or rectal cancer. Chemoradiotherapy for rectal cancer (as a component of curative treatment) is acceptable. NOTE: Patients who achieve a clinical complete response and opt for a non-operative approach to their primary tumor management are not eligible.

  * Patients must be ctDNA-positive by an assay run in any CLIA-certified lab obtained within 2-12 weeks following completion of definitive all curative therapy for colorectal cancer.
  * Tumor status of microsatellite stability (MSS) or Proficient mismatch repair (pMMR) is confirmed through a standard of care assay through a CLIA-certified lab.
* At the time of study entry, blood counts performed within 28 days prior to study entry must meet the following criteria:

  * ANC must be greater than or equal to (≥) 1000/mm3,
  * Platelet count must be ≥ to 80,000/mm3; and
  * Hemoglobin must be ≥ 8 g/dL. (Note: transfusions may be used to correct hemoglobin for patients experiencing anemia from therapy who otherwise would be eligible for the study.)
  * Albumin greater than (>) 3.0 g/dL.
* The following criteria for evidence of adequate hepatic function performed within 28 days prior to study entry must be met:

  * Total bilirubin less than or equal to (≤) 1.5 x ULN
  * AST and ALT must be ≤ 3.0 x ULN for the lab. (Note: In patients with elevated ALT or AST, the values must be stable for at least 2 weeks and with no evidence of biliary obstruction on imaging.)
* Creatinine must be ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 40mL/min.
* All prior chemotherapy toxicities (excluding alopecia, amenorrhea, and peripheral neuropathy) must be less than (<) Grade 2 at the time study therapy is to begin unless AE(s) are clinically stable on supportive therapy.
* Patients must have no evidence of opportunistic infections.
* Patients of childbearing potential must have a negative pregnancy per institutional policies prior to receiving the first dose of study therapy.
* Male and female patients with reproductive potential must agree to use accepted effective methods of contraception while receiving study therapy and for at least 180 days (6 months) after the completion of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria:

* Colon cancer other than adenocarcinoma, e.g., sarcoma, lymphoma, carcinoid.
* Patients with MSI-high (dMMR) tumors.
* Use and/or receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, targeted therapy, biologic therapy, monoclonal anti-bodies) or radiation therapy within 4 weeks prior to receiving first dose of study therapy or associated with immune-mediated adverse events (imAEs) that were Grade ≥1 within 90 days prior to the first dose of study therapy or associated with toxicity that resulted in discontinuation of the immune-modulating agent.
* History of active or latent tuberculosis (TB) infection. If the presence of TB (active or latent) is established, then treatment for TB must be completed according to local guidelines prior to the screening.
* Active untreated or uncontrolled systemic fungal, bacterial, or viral infections, or active infection requiring systemic anti-infectious therapy.
* Current or history of systemic autoimmune disease requiring systemic immunosuppressive therapy will not be allowed. Note: the following will not be exclusionary: 1) the presence of laboratory evidence of autoimmune disease (e.g., positive antinuclear antibody titer or lupus anticoagulant) without associated symptoms; 2) clinical evidence of vitiligo or other forms of depigmenting illness; 3) mild autoimmunity not impacting the function of major organs (e.g., controlled Hashimoto thyroiditis, limited psoriasis), Type I diabetes.
* Patients will be excluded if they are on systemic steroid therapy that cannot be discontinued (except for the use of prednisone or equivalent <0.125mg/kg/day as replacement therapy). Inhaled or topical steroids are permitted.
* Receipt of live attenuated vaccination within 30 days prior to study entry.
* Known active or chronic hepatitis B virus (HBV) or hepatitis C virus (HCB) infections.

Note: Patients with a history of hepatitis C virus (HCV) infection must have been treated and with confirmation of cure, can be eligible.

* History of allogeneic organ or bone marrow transplantation.
* Any of the following cardiovascular conditions:

  * Documented NYHA Class II, III or IV congestive heart failure,
  * History of myocardial infarction (MI), angina pectoris, or coronary artery bypass graft (CABG) within 6 months prior to starting study treatment
  * Transient ischemic attack (TIA) or stroke within 1 year.
  * History of myocarditis
  * Troponin T (TnT) or troponin I (TnI) > 2x institutional ULN at baseline. Patients with TnT or TnI levels between > 1 to 2x ULN are permitted if repeat levels within 24 hours are ≤ 1x ULN. If TnT or TnI levels are > 1 to 2x ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment by the investigator based on medical judgement in the patient's best interest.
* Active, documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* Major surgical procedure within 28 days prior to study entry.
* Other malignancies: unless the patient is considered disease-free and has completed therapy for the malignancy greater than or equal to 36 months prior to study entry. Patients with the following cancers are eligible if diagnosed and definitively treated within the past 12 months: carcinoma in situ of the cervix, and basal cell and squamous cell carcinoma of the skin. Other in situ neoplasms will be reviewed by the Protocol Officer and/or Protocol Chair.
* Psychiatric or addictive disorders or other conditions that in the opinion of the investigator would preclude the patient from meeting the study requirements or interfering with interpretation of study results.
* Pregnancy or lactation at the time of study entry.
* Use of any investigational agent within 28 days prior to the first dose of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Clearance of cDNA | From enrollment to 12 weeks
  To determine the proportion of patients who convert from ctDNA positive at baseline (a condition of eligibility) to ctDNA negative at the 12 week timepoint

SECONDARY OUTCOMES:
Sustainability of clearance of ctDNA | From enrollment to 12 months
  In the subset of patients who did clear ctDNA by 12 weeks (see the primary outcome), to determine the proportion of patients that remain ctDNA-negative at 12 months from trial enrollment.
Sustainability of clearance of ctDNA | From enrollment to 18 months
  In the subset of patients who did clear ctDNA by 12 weeks (see the primary outcome), to determine the proportion of patients that remain ctDNA-negative at 18 months from trial enrollment.
Kinetics of ctDNA clearance in MRD in patients crossing over from cemiplimab monotherapy | From crossover to 18 months after enrollment
  In the subset of patients who cross over from the cemiplimab monotherapy arm, to determine the proportion of patients who convert to ctDNA negative at 12 weeks after crossover, and at 12 and 18 months after study entry.
MRD Response by quantitative ctDNA | From enrollment up to 3 years
  To determine the percentage of patients whose MRD show a response to the trial regimen, including both clearance of ctDNA and partial ctDNA quantitative response defined as decrease in the burden of quantitative ctDNA from baseline.
Recurrence-free survival (RFS) | From enrollment up to 3 years
  To determine time to imaging recurrence following initiation of study therapy through follow-up
Safety [Will be performed on the ITT population] | During study therapy and up to 60 days post therapy, approximately up to 425 days
  To describe the adverse events observed for each arm of the study according to the CTCAE version 5.0
Number of participants with Toxicity [Will be performed on the ITT population] | During study therapy and up to 60 days post therapy, approximately up to 425 days
  To describe the reasons for early termination of therapy